CLINICAL TRIAL: NCT07291388
Title: Effectiveness of Retrolaminar Block in Reducing Postoperative Opioid Consumption in Patients Undergoing Lumbar Spine Fusion With Multimodal Analgesia
Brief Title: Effectiveness of Retrolaminar Block in Lumbar Spine Fusion With Multimodal Analgesia
Acronym: RBLUF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 241022008
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-08

CONDITIONS: Acute Pain; Anesthesia; Lumbar Spine Disease
Keywords: acute pain; retrolaminar block; regional anesthesia; lumbar arthrodesis
MeSH Terms: conditions — Acute Pain; Spinal Diseases; Ankylosis

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, two-group clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Due to the nature of the intervention, both patients and healthcare personnel involved in the intraoperative and postoperative care of the patients will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrolaminar block (Experimental): Participants received retrolaminar block with 0.25% Bupivacaine (20 ml) plus epinephrine (5 mcg/ml), on both sides of the vertebral lamina, and a subcutaneous injection in the area of the surgical incision with 20 ml of the same concentration and dose used previously.
  Interventions: Procedure: retrolaminar block
- Sham block (Sham Comparator): Participants received a retrolaminar sham block with 0.9% saline solution (20 ml), on both sides of the vertebra lamina, and a subcutaneous injection in the area of the surgical incision with 20 ml of the same concentration and dose used previously.
  Interventions: Procedure: Sham block

INTERVENTIONS:
Procedure: retrolaminar block — Retrolaminar block with bupivacaine and epinephrine on both sides of the vertebral lamina, and subcutaneous injection in the area of the surgical incision.
  Arms: Retrolaminar block
Procedure: Sham block — Sham block in the retrolaminar area with saline solution on both sides of the vertebral lamina, and subcutaneous injection in the area of the surgical incision.
  Arms: Sham block

SUMMARY:
This randomized, blinded, controlled clinical trial aims to evaluate the effectiveness of ultrasound-guided retrolaminar block in reducing postoperative opioid consumption in patients undergoing lumbar spine fusion surgery under multimodal analgesia.

The participants will:

* Be randomly assigned in a 1:1 ratio to receive either a retrolaminar block with 0.25% bupivacaine plus epinephrine or a sham block (normal saline) prior to surgical incision.
* Receive standardized multimodal analgesia.
* Have follow-up by the Acute Pain Unit during the first 3 days, to assess opioid consumption (morphine) in 24 hours, pain intensity measured by Numeric Rating Scale, quality of recovery assessed by the QoR-15 questionnaire, intraoperative blood loss, and postoperative complications.

DETAILED DESCRIPTION:
After obtaining approval from the institutional CEC-CCSS and prospective registration of the study at clinicaltrials.org, the investigators will recruit patients who meet the inclusion criteria and provide written consent.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years, scheduled for lumbar spine fusion surgery by a trauma team
* American Society of Anesthesiologists (ASA) Classification I-III
* Willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

* History of chronic use of strong or weak opioids for more than 3 months.
* Diagnosis of chronic pain and treatment by a pain management team.
* ASA score greater than or equal to 4.
* Patients with prior lumbar spine surgery. Spinal instrumentation at the surgical site.
* Estimated creatinine clearance less than 60 ml/min.
* Coagulation disorder or abnormal coagulation tests.
* Infection at the surgical site.
* Weight less than 50 kg.
* Altered mental status that prevents reliable evaluation.
* Allergy to local anesthetics or analgesic drugs used in the study.
* Patients with contraindications to peripheral nerve blocks.
* Lumbar spine fixation due to oncologic disease or acute trauma.
* Use of intraoperative neuromonitoring and TIVA.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption during the first 24 hours postoperative | Daily consumption during the first 24 hours
  To assess rescue opioid consumption, expressed as morphine equivalents, during the first 24 hours postoperative.

SECONDARY OUTCOMES:
Daily Numeric Rating Score (NRS) during the first 3 postoperative days | Daily NRS during the first 3 postoperative days
  The NRS (Numeric Rating Scale) is commonly used to assess pain intensity. Its minimum score is 0, indicating no pain, and its maximum score is 10, indicating the worst pain imaginable. This scale is simple and allows patients to rate their pain using a number from 0 to 10. The objective is to assess the intensity of acute postoperative pain, expressed as NRS, during the first 3 postoperative days.
Daily score on the "Quality of Recovery-15" (QoR-15) scale during the first 3 postoperative days. | Preoperative score and daily score during the first 3 postoperative days
  The QoR-15 is a validated instrument in the literature that assesses the quality of recovery in patients after surgery. It is a multidimensional measurement tool that allows healthcare professionals to gain an overview of the patient's well-being during the postoperative period. The questionnaire consists of 15 items, covering 5 dimensions: Physical Comfort, Physical Independence, Emotional Support, Psychological Well-being, and Satisfaction with Recovery. The minimum score on the scale is 0 points, and the maximum score is 150 points. This range is obtained by summing the scores of the different categories evaluated in the QoR-15 scale, where a higher score indicates a better quality of postoperative recovery.
bleeding and transfusions | Intraoperative and during the first 3 days
  Subjective assessment of total intraoperative bleeding (mild, moderate, severe), blood in collectors, number of compresses with blood, hematocrit variations at 24 hours after the procedure and need for transfusion in the perioperative period.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Machado GC, Ferreira PH, Harris IA, Pinheiro MB, Koes BW, van Tulder M, Rzewuska M, Maher CG, Ferreira ML. Effectiveness of surgery for lumbar spinal stenosis: a systematic review and meta-analysis. PLoS One. 2015 Mar 30;10(3):e0122800. doi: 10.1371/journal.pone.0122800. eCollection 2015. PMID 25822730
- [Background] Pepper CG, Mikhaeil JS, Khan JS. Perioperative Regional Anesthesia on Persistent Opioid Use and Chronic Pain after Noncardiac Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Anesth Analg. 2024 Oct 1;139(4):711-722. doi: 10.1213/ANE.0000000000006947. Epub 2024 Sep 4. PMID 39231035
- [Background] Kaye AD, Kandregula S, Kosty J, Sin A, Guthikonda B, Ghali GE, Craig MK, Pham AD, Reed DS, Gennuso SA, Reynolds RM, Ehrhardt KP, Cornett EM, Urman RD. Chronic pain and substance abuse disorders: Preoperative assessment and optimization strategies. Best Pract Res Clin Anaesthesiol. 2020 Jun;34(2):255-267. doi: 10.1016/j.bpa.2020.04.014. Epub 2020 May 7. PMID 32711832
- [Background] Garg B, Ahuja K, Sharan AD. Regional Anesthesia for Spine Surgery. J Am Acad Orthop Surg. 2022 Sep 1;30(17):809-819. doi: 10.5435/JAAOS-D-22-00101. Epub 2022 May 25. PMID 35617645
- [Background] Voscopoulos C, Palaniappan D, Zeballos J, Ko H, Janfaza D, Vlassakov K. The ultrasound-guided retrolaminar block. Can J Anaesth. 2013 Sep;60(9):888-95. doi: 10.1007/s12630-013-9983-x. PMID 23797663
- [Background] Onishi E, Toda N, Kameyama Y, Yamauchi M. Comparison of Clinical Efficacy and Anatomical Investigation between Retrolaminar Block and Erector Spinae Plane Block. Biomed Res Int. 2019 Mar 28;2019:2578396. doi: 10.1155/2019/2578396. eCollection 2019. PMID 31032339
- [Background] Karmakar MK, Sivakumar RK, Sheah K, Pangthipampai P, Lonnqvist PA. Quest for the Elusive Mechanism of Action for the Thoracic Paraspinal Nerve Block Techniques. Are We Ignoring the Anatomy of the "Retro Superior Costotransverse Ligament Space?". Anesth Analg. 2023 Aug 1;137(2):458-465. doi: 10.1213/ANE.0000000000006462. Epub 2023 Jul 14. No abstract available. PMID 37450909
- [Background] Peker K, Aydin G, Gencay I, Saracoglu AG, Sahin AT, Ogden M, Peker SA. The effect of preemptive retrolaminar block on lumbar spinal decompression surgery. Eur Spine J. 2024 Nov;33(11):4253-4261. doi: 10.1007/s00586-024-08219-4. Epub 2024 Jun 17. PMID 38886235
- [Background] Schnabel A, Yahiaoui-Doktor M, Meissner W, Zahn PK, Pogatzki-Zahn EM. Predicting poor postoperative acute pain outcome in adults: an international, multicentre database analysis of risk factors in 50,005 patients. Pain Rep. 2020 Jul 27;5(4):e831. doi: 10.1097/PR9.0000000000000831. eCollection 2020 Jul-Aug. PMID 32766467
- [Background] Morales-Ariza V, Loaiza-Aldean Y, de Miguel M, Pena-Navarro M, Martinez-Silva O, Gonzalez-Tallada A, Manrique-Munoz S, de Nadal M. Validation and cross-cultural adaptation of the postoperative quality of recovery 15 (QoR-15) questionnaire for Spanish-speaking patients: A prospective cohort study. Am J Surg. 2023 Apr;225(4):740-747. doi: 10.1016/j.amjsurg.2022.11.009. Epub 2022 Nov 17. PMID 36414472
- [Background] Chazapis M, Walker EM, Rooms MA, Kamming D, Moonesinghe SR. Measuring quality of recovery-15 after day case surgery. Br J Anaesth. 2016 Feb;116(2):241-8. doi: 10.1093/bja/aev413. PMID 26787793
- [Background] Kaciroglu A, Ekinci M, Gurbuz H, Ulusoy E, Ekici MA, Dogan O, Golboyu BE, Alver S, Ciftci B. Surgical vs ultrasound-guided lumbar erector spinae plane block for pain management following lumbar spinal fusion surgery. Eur Spine J. 2024 Jul;33(7):2630-2636. doi: 10.1007/s00586-024-08347-x. Epub 2024 Jun 4. PMID 38834814